CLINICAL TRIAL: NCT03018782
Title: The Implementation of a Novel Pain-screening Tool in the Diagnoses of Pain Symptoms and Syndromes in Refugee Survivors of Torture
Brief Title: Pain Screening in Refugee Survivors of Torture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1608017472
Record Dates: First submitted 2016-12-17; First posted 2017-01-12 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief Pain Inventory Short Form (Other): Completes the Brief Pain Inventory Short Form
  Interventions: Other: Brief Pain Inventory Short Form

INTERVENTIONS:
Other: Brief Pain Inventory Short Form — Brief Pain Inventory Short Form

SUMMARY:
The investigators are evaluating refugee torture survivors who are receiving services at the Weill Cornell Center for Human Rights. There are two research questions in this study: if the current standard of care results in the under or missed diagnosis of pain and pain syndromes, and if a validated pain screening tool can supplement the current standard protocol used in the assessments of survivors of torture.

DETAILED DESCRIPTION:
The research plan consists of three components:

1. The Weill Cornell Center for Human Rights will coordinate with the research team regarding eligible subjects.
2. Researchers will contact potential subjects utilizing interpreter services.
3. Interested participants will be scheduled for an appointment for an examination by a pain physician and to complete the Brief Pain Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from any country over the age of 18
* refugees receiving services from the Weill Cornell Center for Human Rights

Exclusion Criteria:

* Have not experienced torture
* Subjects whose representative does not believe that they are a good candidate for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with chronic pain or pain syndromes as assessed by a non-invasive pain evaluation conducted by a pain physician | Day 1
  Evaluate whether or not current standard protocols for the assessment of survivors of torture result in under or missed diagnosis of pain and pain syndromes that are identifiable by a pain specialist physician

SECONDARY OUTCOMES:
Number of participants with chronic pain or pain syndromes as assessed by the Brief Pain Inventory (BPI) Short Form | Day 1
  Evaluate whether or not a validated pain screening tool can supplement the current standard protocols used in the assessment of survivors of torture.

CONTACTS AND LOCATIONS:
Overall Officials: Gunisha Kaur, MD, Principal Investigator — Weill Medical College of Cornell University; Eliana Weinstein, BS, Study Director — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Derived] Kaur G, Weinberg R, Milewski AR, Huynh S, Mauer E, Hemmings HC Jr, Pryor KO. Chronic pain diagnosis in refugee torture survivors: A prospective, blinded diagnostic accuracy study. PLoS Med. 2020 Jun 5;17(6):e1003108. doi: 10.1371/journal.pmed.1003108. eCollection 2020 Jun. PMID 32502219